CLINICAL TRIAL: NCT02739776
Title: Infrared Thermographic Imaging for Early Assessment of Epidural Block Success in Obstetric Anesthesia
Brief Title: Thermographic Imaging in Epidural Anesthesia
Status: Withdrawn | Type: Observational
Why Stopped: incomplete information
Sponsor: Cook County Health (Other Government)
Responsible Party: Principal Investigator, Pamela Gonzalez Sr Director Clinical Research Office, Dir Clinical Research, Cook County Health
Other Study IDs: IRB# 16-012
Record Dates: First submitted 2016-03-29; First posted 2016-04-15 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Epidural Blockade

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Pt receiving standard Epidural block care for vaginal delivery
  Interventions: Device: Thermographic imaging

INTERVENTIONS:
Device: Thermographic imaging — Using infrared-recording camera will obtain thermographic images of the lower extremities before and after the epidural blockade

SUMMARY:
The purpose of this study is to describe infrared thermographic imaging as a tool for the assessment of epidural block in obstetrics patients

DETAILED DESCRIPTION:
Patients will recive standard anesthesia care for epidural placement and additionally, thermographic imaging will be obtained at baseline and up to 30 min after the epidural blockade is performed.

ELIGIBILITY:
Inclusion Criteria:

* Parturients in active labor requesting epidural anesthesia for normal vaginal delivery

Exclusion Criteria:

* Patients with lower extremity skin disorders like active infections like cellulitis, ,dermatitis, psoriasis or connective tissue disorders like scleroderma or Raynaud's phenomenon
* Patients with diagnosed peripheral vascular disease ,venous stasis , deep venous thrombosis.
* Patients with Severe preeclampsia with significant lower extremity edema
* Patient on vasoactive agents like vasodilators, calcium channels blockers.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parturients in active labor, older than18 year of age, requesting epidural anesthesia for normal vaginal delivery
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2017-11-17 (Actual); Study Completion 2017-11-17 (Actual)

PRIMARY OUTCOMES:
Change in temperature in the lower extremities | at baseline, 5 min before the epidural blockade, during and up to 30 minutes after performing the epidural blockade
  thermographic images of the lower extremities will be obtained and analyzed for thermography patterns.

SECONDARY OUTCOMES:
Successful epidural blockade | up to 30 min after performing the epidural block
  adequate sensory level, pain control, motor blockade as evaluated by care provider
Epidural blockade failure | Up to 30 min after performing the epidural block
  Failure of the epidural block to adequately control pain, unilateral blockade, optimal sensory level, inadequate motor blockade
Requirement for Epidural catheter manipulation or replacement | Up to 30 min after performing the epidural block

OTHER OUTCOMES:
Peri-procedural Complications | participants will be followed for the duration of anesthesia and after the procedure, an expected average of 12 hours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galvin EM, Niehof S, Medina HJ, Zijlstra FJ, van Bommel J, Klein J, Verbrugge SJ. Thermographic temperature measurement compared with pinprick and cold sensation in predicting the effectiveness of regional blocks. Anesth Analg. 2006 Feb;102(2):598-604. doi: 10.1213/01.ane.0000189556.49429.16. PMID 16428569
- [Background] Kim YC, Bahk JH, Lee SC, Lee YW. Infrared thermographic imaging in the assessment of successful block on lumbar sympathetic ganglion. Yonsei Med J. 2003 Feb;44(1):119-24. doi: 10.3349/ymj.2003.44.1.119. PMID 12619184
- [Background] Asghar S, Lundstrom LH, Bjerregaard LS, Lange KH. Ultrasound-guided lateral infraclavicular block evaluated by infrared thermography and distal skin temperature. Acta Anaesthesiol Scand. 2014 Aug;58(7):867-74. doi: 10.1111/aas.12351. Epub 2014 Jun 12. PMID 24924688